CLINICAL TRIAL: NCT03785717
Title: Horizontal Guide Bone Regeneration With or Without Shock Waves: a Randomized Clinical Trial
Brief Title: Horizontal Ridge Augmentation in Mandible Usign ROG + ESWT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad El Bosque, Bogotá (Other)
Collaborators: Gloria Lafaurie (Unknown); Carlos Leal (Unknown)
Responsible Party: Principal Investigator, Yamil Lesmes, DDS, MSc candidate, Universidad El Bosque, Bogotá
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PCI2015-8351
Record Dates: First submitted 2018-03-02; First posted 2018-12-24 (Actual); Last update posted 2018-12-24 (Actual); Status verified 2018-12

CONDITIONS: Bone Regeneration
Keywords: shock wave therapy (SWT or ESWT); Guided bone regeneration (GBR); horizontal ridge augmentation
MeSH Terms: conditions — Ciliary Dyskinesia, Primary, 13

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ROG only (Active Comparator): cancellous (1-2 mm) & cortical (250-1000 mm) bone allograft and pericardium membrane without extracorporeal shockwave therapy
  Interventions: Procedure: ROG; Procedure: ROG & ESWT
- ROG & ESWT (Active Comparator): cancellous 1-2mm & cortical 250-1000mm Bonegrafts and membrane with extracorporeal shockwave therapy
  Interventions: Procedure: ROG; Procedure: ROG & ESWT

INTERVENTIONS:
Procedure: ROG — Bone width augmentation using bone grafting and membrane non cross linking.
Procedure: ROG & ESWT — Before the bone width augmentation using bone grafting and membrane non cross linking, the patient was received ESWT (Extracorporeal shockwave therapy).

SUMMARY:
Guided bone regeneration (GBR) has been the most frequently used option to treat bone ridge deficiencies, allowing to restore such defects in order to place bone-integrated dental implants. A few reports exist in the literature about the augmentation of mandibular horizontal ridge defects before implant placement. Published studies show a large variability of reported results regarding horizontal bone augmentation. This can be due to the use of different types of membranes and bone graft materials or a combination thereof. Likewise, an important percentage of graft reabsorption is reported. Although this technique is very much used, an important number of cases must be re-treated or require placing bone graft during implant installation surgery. Techniques are required in order to improve vascularization of the grafts during GBR technique with the aim to improve their clinical success. Recent studies show great interest on the application of shock waves in oral diseases associated to infection and bone loss. The shock waves are acoustic waves that have effects on human biological tissues, stimulating the neo-angiogenesis and the development of a hyper cellularity, showing repairing characteristics on tissues, and starting regenerative processes as a result of metabolism improvement and the increase of local circulation. The extra corporeal shock waves can activate the osteoblasts and their precursors and they have been widely used in orthopaedics for repairing bone fractures. Several clinical studies have shown the effectiveness and safety of shock wave therapy in myocardial revascularization, lithotripsy, cellulitis, volar fasciitis, osteonecrosis, bone fractures, and complicated injuries of soft tissues. No clinical studies exist that assess its effect on guided bone regeneration. The evidence related to the positive effects of the use of shock waves on bone regeneration suggests this treatment as a novelty and a promising therapy that combined with the GBR technique for the treatment of horizontal defects could have an important impact on the potentialization of its clinical effectiveness.

DETAILED DESCRIPTION:
General Objective:

Assessing the efficacy of horizontal augmentation and percentage of reabsorption of bone graft material in the technique of guided bone regeneration (GBR), combined with the shock wave therapy (SWT) in the horizontal bone reconstruction of mandibular alveolar ridges.

Type of study:

Triple blind randomized clinical trial

Population and sample:

Twenty six patients of university and private clinical practice, who require augmentation of horizontal ridge in the mandible for back placing of an implant, and their compliance with inclusion and exclusion criteria, will be assessed.

Type of analysis:

Central trend and dispersion (medium and standard deviation) measurements will be obtained. Type of data distribution using Shapiro Wilk.

t-student test between no related groups for assessing bone augmentation. t-paired test between related groups for assessing pre and post treatment within the same group.

t test for proportion difference, in order to assess the percentage of reabsorption of bone graft, bone density, bone quality, within a same group.

Fisher, group comparison.

A multiple linear regression model will be developed in order to establish if the difference among groups is influenced by the initial width of the ridge and the thickness of the soft tissue.

In case of not following a normal distribution, no parametrical tests for related and no related groups and logistic regression, will be used.

The frequencies of adverse effects in each group will be obtained, and compared to the Chi2 test or the Fisher exact test.

All the analyses will be made with significance level of 5% (p< 0.05).

Effect measurements: Relative Risk (RR), Attributable Risk Reduction (ARR), and Necessary Number to be Treated (NNT). The augmentation of horizontal volume that allows the installation of a ≥4.1 mm implant will be taken as cutting point reference of clinical success.

Expected Results:

* Establishing the effect of the shock wave therapy, in combination with guided bone regeneration, on the improvement of bone augmentation and the decrease of bone graft reabsorption.
* Establishing the effect of shock wave therapy, in combination with guided bone regeneration, on the improvement of bone quality and density, as well as on decreasing the adverse effects.
* Acquiring new knowledge in the area of bone reconstruction.
* Presentation of results in local and international congresses.
* Formation of human resource; mastery graduation paper on Dentistry Science Master.

ELIGIBILITY:
Inclusion Criteria:

* Patients who agree to participate in the study and sign informed consent
* Partial mandibular edentulism requiring at least two teeth to be replaced with osseointegrated implants
* Patient with alveolar ridge thickness of ≤4mm, evaluated by CBCT
* Vertical bone availability of 9mm to anatomical structure such as a chin or dental canal that allows a short implant placement of 8mm at the end of the study.
* Extractions performed ≥ 6 months
* Elderly patients between 35 and 65 years old
* Patients without current disease or with chronic pathologies in medical control that does not affect the healing processes such as: controlled hypertension, controlled hypothyroidism, controlled hypercholesterolemia
* Evaluated by anamnesis and laboratory tests that rule out processes of immunosuppression, glycemia and coagulation disorders hypercholesterolemia
* No smoking

Exclusion Criteria:

* Diabetes
* Immunosuppressive drugs
* Anti-coagulated or with dual anti-platelet aggregation
* Therapy with bisphosphonates
* Hormone replacement therapy
* Patient with a history of radiotherapy of the head and neck
* Pregnant women or nursing
* Permanent consumption of NSAIDs and corticosteroids
* Prolonged antibiotic therapy in the last 6 months

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-12-11 (Actual); Study Completion 2018-12-20 (Actual)

PRIMARY OUTCOMES:
Change in Bone width (in mm), as assessed using (CBCT) on a partially edentulous patients after ROG+ESWT. | Patients will be assessed prior the ROG, two weeks after ROG, and 6 months after ROG in order to determinate actual situation, the situation after the ROG placement and the reabsorption of ROG material.
  Using specialized software in dental implantology, measurements are taken in the tomographies taken of each volunteer patient, in order to determine the increase in bone volume in the intervention, and its reabsorption after the healing process.

CONTACTS AND LOCATIONS:
Overall Officials: Yamil Lesmes, Principal Investigator — Universidad El Bosque
Locations (1):
- Yamil Lesmes, Bogotá, Colombia

IPD SHARING:
Plan to Share IPD: Undecided